CLINICAL TRIAL: NCT05294666
Title: Evaluation of Efficacy, Safety and Tolerability of 0.05% Cyclosporine and 0.1% Tacrolimus Eye Drops in the Treatment of Chronic Ocular Graft-versus-host Disease
Brief Title: Evaluation of 0.05% CsA and 0.1% FK506 Eye Drops in Ocular GVHD Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99304
Record Dates: First submitted 2022-02-07; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-01

CONDITIONS: Graft Versus Host Disease in Eye
Keywords: ocular graft-versus-host disease; dry eye; cyclosporine; tacrolimus; prospective study
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cyclosporine group (Experimental): The chronic ocular GVHD patients in cyclosporine group received local 0.05% cyclosporine 4 times/day for 3 months, and then changed to 0.05% cyclosporine for 2 times/day for 3 months
  Interventions: Drug: Cyclosporine
- tacrolimus group (Experimental): The chronic ocular GVHD patients in tacrolimus group received local 0.05% tacrolimus 2 times/day for 3 months, and then changed to 0.05% cyclosporine for 2 times/day for 3 months
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: Cyclosporine — The chronic ocular GVHD patients in cyclosporine group received local 0.05% cyclosporine 4 times/day for 3 months, and then changed to 0.05% cyclosporine for 2 times/day for 3 months
  Other Names: CsA
  Arms: cyclosporine group
Drug: tacrolimus — The chronic ocular GVHD patients in tacrolimus group received local 0.05% tacrolimus 2 times/day for 3 months, and then changed to 0.05% cyclosporine for 2 times/day for 3 months
  Other Names: FK506
  Arms: tacrolimus group

SUMMARY:
It is planned to explore the efficacy and safety of local 0.05% cyclosporine eye drops in the treatment of chronic graft-versus-host eye disease. Through the comparative study with 0.1% tacrolimus eye drops, to clarify the short-term and long-term efficacy of 0.05% CSA in these patients, and to explore the benefits of long-term maintenance of local cyclosporine to patients.

DETAILED DESCRIPTION:
Chronic graft-versus-host disease (GVHD) is a common and serious complication after allogeneic hematopoietic stem cell transplantation. Its clinical presentation is similar to that of an autoimmune disease and can affect many organs, including the skin, liver, gastrointestinal tract, lungs and eyes. Ocular GVHD occurs in 30-60% of patients undergoing hematopoietic stem cell transplantation and 60-90% of patients with other systemic GVHD. Chronic ocular GVHD usually occurs 9-24 months after hematopoietic stem cell transplantation and mainly affects the cornea, conjunctiva, lacrimal gland, eyelid and meibomian gland, and leads to inflammation and fibrosis of these tissues. The characteristic manifestations of chronic GVHD include dry keratoconjunctivitis, cicatric conjunctivitis, punctate keratopathy, corneal ulcer and perforation. Severe dry eye is the most common manifestation of ocular GVHD. Patients have burning sensation, foreign body sensation, photophobia, dry eye, itching and other symptoms. This is associated with reduced tear secretion due to damage to the lacrimal gland as well as with goblet cell loss and tear film instability due to meibomian gland dysfunction. Chronic eye GVHD has the potential to cause severe visual impairment and significantly reduce the patient's quality of life. The principle of topical treatment of ocular GVHD is to lubricate the ocular surface, reduce ocular surface inflammation, prevent tear evaporation, and promote epithelial repair. Specific local treatment options include glucocorticoids, immunosuppressants, growth factors and artificial tears. Local glucocorticoids are the first-line treatment at the present stage, but the side effects of hormone therapy are relatively large. Long-term use can lead to damaged epithelial formation, thinning of the cornea, increased intraocular pressure, cataract, infectious keratitis, etc. Therefore, it is necessary to closely monitor the treatment period and minimize the use time. At present, the most commonly used topical immunosuppressants are tacrolimus (FK506) and cyclosporine (CsA). Both belong to calcineurin inhibitors, which can inhibit the activation of calcium-dependent T cells, thus exerting immunosuppressive effect. 0.05% CsA is an eye drop mainly used for the treatment of moderate and severe dry eye, with good therapeutic effect and tolerability [18-23], but slow onset of effect. In the treatment of patients with chronic ocular GVHD, previous studies have shown that cyclosporine eye drops can improve patients' dry eye symptoms, reduce corneal fluorescence staining, and increase tear film rupture time. However, the number of clinical studies on the treatment of chronic ocular GVHD with 0.05% CsA eye drops is limited, with a small number of patients enrolled and relatively short follow-up time. The immunosuppressive effect of tacrolimus is significantly higher than cyclosporine, which is 100 times higher than reported in literature. Therefore, tacrolimus is mainly used for the treatment of rejection after corneal transplantation and immune-related ocular surface diseases. What is the efficacy and tolerability of such a powerful immunosuppressant in treating GVHD? There are few literature reports, but long-term ocular application can reduce local immunity and increase the risk of local infection. At the same time, tacrolimus is very irritating, and some patients cannot tolerate it and choose to stop using the drug. At present, there is still a lack of clinical evidence to compare the efficacy of cyclosporine and tacrolimus eye drops in patients with chronic ocular GVHD. Therefore, by comparing the effectiveness, safety and tolerance of 0.05% CsA eye drops and 0.1% tacrolimus eye drops in the treatment of chronic eye graft-versus host eye disease, this study aims to explore a reasonable treatment plan for chronic eye GVHD and provide theoretical basis for clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as chronic ocular GVHD
* Did not receive eye local immunosuppressive therapy
* Non pregnant patients

Exclusion Criteria:

* Have a history of eye surgery in the past six months
* Suffering from other eye diseases (autoimmune diseases, glaucoma, serious infection, retinopathy, allergy, cataract, eye trauma, etc.)
* Hormones or immunosuppressants were used before enrollment

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
visual acuity | Within 4 hours of initial enrollment
  visual acuity
visual acuity | At the first month of enrollment
  visual acuity
visual acuity | At the third month of enrollment
  visual acuity
visual acuity | At the sixth month of enrollment
  visual acuity
Intraocular pressure | Within 4 hours of initial enrollment
  Intraocular pressure
Intraocular pressure | At the first month of enrollment
  Intraocular pressure
Intraocular pressure | At the third month of enrollment
  Intraocular pressure
Intraocular pressure | At the sixth month of enrollment
  Intraocular pressure
Ocular Surface Disease Index | Within 4 hours of initial enrollment
  Ocular Surface Disease Index
Ocular Surface Disease Index | At the first month of enrollment
  Ocular Surface Disease Index
Ocular Surface Disease Index | At the third month of enrollment
  Ocular Surface Disease Index
Ocular Surface Disease Index | At the sixth month of enrollment
  Ocular Surface Disease Index
Corneal fluorescein staining | Within 4 hours of initial enrollment
  Corneal fluorescein staining
Corneal fluorescein staining | At the first month of enrollment
  Corneal fluorescein staining
Corneal fluorescein staining | At the third month of enrollment
  Corneal fluorescein staining
Corneal fluorescein staining | At the sixth month of enrollment
  Corneal fluorescein staining
Tear break-up time | Within 4 hours of initial enrollment
  Tear break-up time
Tear break-up time | At the first month of enrollment
  Tear break-up time
Tear break-up time | At the third month of enrollment
  Tear break-up time
Tear break-up time | At the sixth month of enrollment
  Tear break-up time

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No